CLINICAL TRIAL: NCT06293261
Title: Multicenter, Prospective, Non-interventional, Observational Study to Confirm the Long-term Efficacy and Safety of Rosuampin Tab. in Patients With Hypertension and Hypercholesterolemia
Status: Completed | Type: Observational
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: YMC043
Record Dates: First submitted 2024-02-28; First posted 2024-03-05 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-11

CONDITIONS: Hypertension; Hypercholesterolemia
Keywords: long-term efficacy and safety of Rusuampin Tab
MeSH Terms: conditions — Hypertension; Hypercholesterolemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Rosuampin 5/5mg (Rosuvastatin 5mg + Amlodipine 5mg)
  Interventions: Drug: Rosuampin 5/5mg, 10/5mg, 20/5mg, 10/10mg
- Rosuampin 10/5mg (Rosuvastatin 10mg + Amlodipine 5mg)
  Interventions: Drug: Rosuampin 5/5mg, 10/5mg, 20/5mg, 10/10mg
- Rosuampin 20/5mg (Rosuvastatin 20mg + Amlodipine 5mg)
  Interventions: Drug: Rosuampin 5/5mg, 10/5mg, 20/5mg, 10/10mg
- Rosuampin 10/10mg (Rosuvastatin
  Interventions: Drug: Rosuampin 5/5mg, 10/5mg, 20/5mg, 10/10mg

INTERVENTIONS:
Drug: Rosuampin 5/5mg, 10/5mg, 20/5mg, 10/10mg — Experimental only, not included active and placebo comparator

SUMMARY:
This study is to confirm the long-term efficacy and safety of Rosuampin Tab. in patients with hypertension and hypercholesterolemia

DETAILED DESCRIPTION:
All treatments, such as drug administration and clinical laboratory tests performed after Rosuampine administration, are performed according to the investigator's medical judgment, and information to be confirmed in this observational study is collected for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 19 years
2. Patients with hypertension and hypercholesterolemia who are receiving Rosuampin medication or need Rosuampin medication according to the medical judgment of the investigator
3. Written informed consent

Exclusion Criteria:

1. Patients with hypersensitivity to components of this drug or other dihydropyridine drugs
2. A woman who is pregnant or likely to be pregnant, a woman of childbearing age who does not use appropriate contraception and a nursing woman
3. a patient with severe liver failure
4. Patients with active liver disease who include continuous serum transaminase elevation of unknown cause or serum transaminase elevation over three times the upper limit of normal
5. a patient with severe aortic valvular stenosis
6. a myopathy patient
7. a cyclosporine co-administered patient
8. a patient with severe renal failure (CLcr, creatinine clearance <30 mL/min)

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with hypertension and hypercholesterolemia who are receiving Rosuampin medication or need Rosuampin medication according to the medical judgment of the investigator
Sampling Method: Probability Sample
Enrollment: 5047 (Actual)
Dates: Start 2020-06-27 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Occurence rate of MACCE(Major Adverse Cardiovascular and Cerebrovascular Events) | Baseline, 12 Months

SECONDARY OUTCOMES:
Change from baseline to 6/12 months in SBP and DBP | Baseline, 6, 12 Months
Percent change from baseline to 6/12 months in Lipid Profile (TC, LDL-C, TG, HDL-C) | Baseline, 6, 12 Months
Change from baseline to 6/12 months in hs-CRP | Baseline, 6, 12 Months
Change from baseline to 6/12 months in Diabetes indicator (Fasting Blood Glucose) | Baseline, 6, 12 Months
Change from baseline to 6/12 months in Diabetes indicator ( HbA1c) | Baseline, 6, 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Moohyun Kim, Principal Investigator — Dong-A University Hospital
Locations (39):
- South Korea (39):
  - Hallym University Sacred Heart Hospital, Anyang-si
  - Dong-A University Hospital, Busan
  - Changwon Fatima Hospital, Changwon
  - Gyeongsang National University Changwon Hospital, Changwon
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Yeungnam University Medical Center, Daegu
  - Daejeon Eulji Medical Center Eulji University, Daejeon
  - Myungji Hospital, Goyang-si
  - Chonnam National University Hospital, Gwangju
  - Chosun University Hospital, Gwangju
  - Bundang Jesaeng General Hospital, Gyeonggi-do
  - Cha University Bundang Medical Center, Gyeonggi-do
  - Hallym University Dongtan Sacred Heart Hospital, Gyeonggi-do
  - Korea University Ansan Hospital, Gyeonggi-do
  - National Health Insurance Service Ilsan Hospital, Gyeonggi-do
  - Samsung Changwon Hospital, Gyeongsang
  - Wonkwang University Hospital, Iksan
  - Dongguk University Ilsan Hospital, Ilsan
  - Inje University Ilsan Paik Hospital, Ilsan
  - Inha University Hospital, Incheon
  - Kwandong University International St.Mary'S Hospital, Incheon
  - Soon Chun Hyang University Hospital Cheonan, Jungbuk
  - Dankook University Hospital, Jungnam
  - Kwangju Veterance Hospital, Kwangju
  - Pusan National University Hospital, Pusan
  - Pusan National University Yangsan Hospital, Pusan
  - Gangnam Severance Hospital, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Ewha Womans University Seoul Hospital, Seoul
  - Hallym University Medical Center, Seoul
  - Kangdong Sacred Heart Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Kyung Hee University Medical Center, Seoul
  - National Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Ulsan University, Ulsan
  - Wonju Severance Christian Hospital, Wŏnju